CLINICAL TRIAL: NCT02968277
Title: LifeWalker Upright Walker Versus Conventional Rollator Walker and Predicate Device
Brief Title: LifeWalker Upright Walker vs. Conventional Rollator Walker and Predicate Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00202634
Record Dates: First submitted 2016-10-25; First posted 2016-11-18 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: No washout period between different arms
Oversight: Data Monitoring Committee: No

ARMS (3):
- Started with Forearm Support Walker (LW Upright) (Experimental): Data collection began with participants using the LifeWalker Upright Walker then using the two remaining walkers in a randomized order
  Interventions: Device: LifeWalker Upright; Device: Predicate Device; Device: Standard Rollator
- Standard Rollator Walker (Control) (Experimental): Data collection began with participants using a conventional standard rollator (SR) walker then using the two remaining walkers in a randomized order
  Interventions: Device: LifeWalker Upright; Device: Predicate Device; Device: Standard Rollator
- Predicate Device (PD) (Experimental): Data collection began with participants using their own rollator walkers then using the two remaining walkers in a randomized order
  Interventions: Device: LifeWalker Upright; Device: Predicate Device; Device: Standard Rollator

INTERVENTIONS:
Device: LifeWalker Upright — LifeWalker (LW) upright walker
Device: Predicate Device — Individual's personal walker
Device: Standard Rollator — A control rollator device

SUMMARY:
The purpose of this project is to evaluate if the LifeWalker Upright walker is improves walking and reports of pain compared to a conventional rollator and predicate walker device.

DETAILED DESCRIPTION:
The LifeWalker Upright is a walker that has been designed to address fall risk, slouching, and user confidence and comfort. The LifeWalker has adjustable armrests and handles that enable users to stand tall and look ahead, providing support and stability that is designed differently than conventional walkers. The LifeWalker Upright's design allows the user to walk within the walker. This allows people to walk inside the walker as opposed to behind the walker.

The purpose of this project is to evaluate if the LifeWalker Upright walker is improves walking and reports of pain compared to a conventional rollator and predicate walker device

Aim 1: Perform in-laboratory training on the Life Walker and testing to compare functional gait outcomes with the Life Walker compared to a conventional rollator and predicate assistive mobility device. We expect that participants will be able to walk longer and will perform more efficiently on measures of gait function when using the Life Walker.

Aim 2: Perform in-laboratory testing to compare self-reported pain with the Life Walker compared to a conventional rollator and predicate assistive mobility device. We expect that participants will report less pain because they will have a more efficient and upright posture when using Life Walker.

Aim 3: Perform in-laboratory testing to compare measures of quality of life with the Life Walker compared to a conventional rollator and predicate mobility device. We expect that participants will report better outcomes on quality of life measures because they will experience better self-esteem due to better mobility when using Life Walker.

Participants will first complete a series of gait testing. Gait testing will include the six minute walk test and the 10 meter walk test. In addition there will be hand and forearm load and grip testing using load sensors. Participants will also be asked to be videotaped during their training sessions. After all the testing is complete, participants will be asked to complete a set of self-report questionnaires. During each device session, participant heart rate, blood pressure and blood oxygenation will be measured. All of these procedures will be repeated with each device.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who use a walker due to back pain or adults (over 18) who use a walker for ambulation.
* Ages from 18 to 89 years old
* Medically stable for therapy

Exclusion Criteria:

* Patient weight exceeds 300 lbs
* Patient height is below 5'0" or exceeds 6'3"
* Inactive, physically unfit to fit into the device.
* Cognitive deficits or visual impairment that would impair their ability to give informed consent or to follow simple instructions during the experiments.
* Mini-Mental State Exam (MMSE) score below 17
* Pregnant women
* Co-morbidity that interferes with the study (e.g. stroke, pace maker placement, severe ischemia cardiac disease, etc.)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jayaraman C, Mummidisetty CK, Loesch A, Kaur S, Hoppe-Ludwig S, Staat M, Jayaraman A. Postural and Metabolic Benefits of Using a Forearm Support Walker in Older Adults With Impairments. Arch Phys Med Rehabil. 2019 Apr;100(4):638-647. doi: 10.1016/j.apmr.2018.10.001. Epub 2018 Oct 24. PMID 30367875

RESULTS

PARTICIPANT FLOW:
Groups:
- Started With Forearm Support Walker (LW Upright): Data collection began with participants using the LifeWalker Upright walker then the other two walkers in a randomized order
- Started With Standard Rollator Walker: Data collection began with participants using a conventional standard rollator (SR) walker then the other two walkers in a randomized order
- Started With Predicate Device (PD): Data collection began with participants using their own rollator walkers then using the two remaining walkers in a randomized order
Period: Overall Study
Arm/Group | Started With Forearm Support Walker (LW Upright) | Started With Standard Rollator Walker | Started With Predicate Device (PD)
Started | 10 | 7 | 13
Completed | 10 | 7 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Started With Standard Rollator Walker: Data collection began with participants using a conventional standard rollator (SR) walker then using the two remaining walkers in a randomized order
- Total: Total of all reporting groups
Arm/Group | Started With Forearm Support Walker (LW Upright) | Started With Standard Rollator Walker | Started With Predicate Device (PD) | Total
Number analyzed (Participants) | 10 | 7 | 13 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 7 | 18
  >=65 years | 4 | 2 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.2) | 61.9 (11.3) | 61.9 (8.4) | 62.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 10 | 24
  Male | 2 | 1 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 13 | 30
Use Walker for Ambulation [Count of Participants; unit: Participants] | 10 | 7 | 13 | 30

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test
Description: The 6 minute walk test is performed as an objective evaluation of functional exercise capacity. The 6minute walk test is easy to administer, well tolerated, and typically reflective of activities of daily living. The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. The number of stops and stumbles will be recorded during the test. This test will be administered while wearing a mask to measure oxygen consumption in addition to blood pressure, heart rate and oxygen saturation.
Time Frame: One testing session
Measure: Mean (Standard Error); unit: meters
Groups:
- Forearm Support Walker (LW Upright): Data collected while participants used the LifeWalker Upright walker.
- Standard Rollator Walker (Control): Data collected while participants used a conventional standard rollator (SR) walker.
- Predicate Device (PD): Data collected while participants used their own rollator walkers.
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator Walker (Control) | Predicate Device (PD)
Number analyzed (Participants) | 30 | 30 | 30
meters | 245.2 (19.1) | 234.7 (18.8) | 233.9 (17.0)

2. Secondary Outcome: 10 Meter Walk Test
Description: Time to walk 10 meters is measured to calculate gait speed.
Time Frame: One testing session
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator Walker (Control) | Predicate Device (PD)
Number analyzed (Participants) | 30 | 30 | 30
meters per second | 1.00 (0.06) | 1.04 (0.07) | 1.01 (0.06)

3. Secondary Outcome: Baseline Modified Falls Efficacy Scale (mFES) Score:
Description: The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling." Subjects answer questions about how confident they are in safely completing various tasks on a scale from 0 to 10, with 10 indicating greater confidence. The score below is the average item-score for the assessment.
Time Frame: Baseline score taken at first session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Started With Forearm Support Walker (LW Upright) | Started With Standard Rollator Walker | Started With Predicate Device (PD)
Number analyzed (Participants) | 10 | 7 | 13
score on a scale | 8.20 (1.6) | 7.47 (0.94) | 6.19 (2.1)

4. Secondary Outcome: Visual Analog Pain Scale (VAS)
Description: The Visual Analog Scale Pain Scale is a measure of perceived pain intensity. It consists of a horizontal line that is 10 centimeters long. On either side of the line is a description of pain- to the left the description will read "No pain," and to the right the description will read "worst pain imaginable." The individual is instructed to mark a point on the continuum which represents his/her pain.
Time Frame: Baseline score taken at first session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Started With Forearm Support Walker (LW Upright) | Started With Standard Rollator Walker | Started With Predicate Device (PD)
Number analyzed (Participants) | 10 | 7 | 13
score on a scale | 4.48 (2.4) | 3.86 (2.2) | 2.77 (2.2)

5. Secondary Outcome: User Functional Rating Scale
Description: Is specifically to assess the user's perception of difficulty in performing the functional tasks when using the different assistive devices. The scale is similar to the patient specific functional scale wherein functional tasks are rated in level of their difficulty from "0" ("inability to perform the task") to "10" ("no difficulty in performing the task.").
Time Frame: One testing session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator Walker (Control) | Predicate Device (PD)
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 7.17 (1.78) | 8.26 (2.07) | 8.58 (1.56)

6. Secondary Outcome: Borg Rate of Perceived Exertion
Description: The Borg Rate of Perceived Exertion is a scale that measures perceived exertion during activity. The minimum score is 6 and the maximum score is 20, with higher values on the scale indicative of higher perceived exertion while completing an activity.
Time Frame: One testing session
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator Walker (Control) | Predicate Device (PD)
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 12 (0.57) | 14.1 (0.64) | 14.1 (0.62)

7. Secondary Outcome: Forearm and Hand Grip
Description: Specialty gloves and load cells will be used to measure to amount of load participants are using when using each device on the hands and also on the forearm. This will be collected during the six-minute walk test.
Time Frame: One testing session
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator Walker (Control) | Predicate Device (PD)
Number analyzed (Participants) | 30 | 30 | 30
kilograms | 4.8 (0.9) | 5.8 (1.05) | 5.7 (0.78)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed, during every data collection session, through study completion, an average of 2 days.
Groups:
- Forearm Support Walker (LW Upright): This arm reflects time during which participants were using the LifeWalker Upright walker
- Standard Rollator (Control): This arm reflects time during which participants were using a standard rollator walker
- Predicate Device (PD): This arm reflects time during which participants were using their own rollator walkers
Arm/Group | Forearm Support Walker (LW Upright) | Standard Rollator (Control) | Predicate Device (PD)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
All assessments were done on level ground surfaces, all tests were done in controlled, clinical environment. Long term effects of using LifeWalker could not be determined in this study. The pathological demographic of the study sample was diverse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02968277/Prot_000.pdf